CLINICAL TRIAL: NCT01665677
Title: Phase II Study of Atorvastatin, Micro-dose Methotrexate and Tacrolimus Administered Only to Transplant Recipients for the Prophylaxis of Acute Graft-versus-host Disease Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Atorvastatin as GVHD Prophylaxis for Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mehdi Hamadani (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Mehdi Hamadani, Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00021090; WVU 011012 (Other: West Virginia); 116837-IRG-09-061-01 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Graft vs Host Disease
Keywords: Graft vs Host Disease; GVHD; Allogeneic hematopoietic stem cell transplantation; HSCT; Atorvastatin
MeSH Terms: conditions — Graft vs Host Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin calcium (Lipitor) (Experimental): Atorvastatin will be administered at a dose of 40 mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning.
  Patients will receive atorvastatin until +180 days or until the patient develops grade II-IV acute GVHD, extensive chronic GVHD, or any grade 3-4 toxicity related to atorvastatin.
  Interventions: Drug: Atorvastatin calcium
- Unrelated Donor (Experimental): Atorvastatin will be administered at a dose of 40 mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning.
  Patients will receive atorvastatin until +180 days or until the patient develops grade II-IV acute GVHD, extensive chronic GVHD, or any grade 3-4 toxicity related to atorvastatin.
  Interventions: Drug: Atorvastatin calcium

INTERVENTIONS:
Drug: Atorvastatin calcium — 40 mg PO daily
  Other Names: Lipitor

SUMMARY:
Hematopoietic stem cell transplantation is a procedure in which a person receives blood forming stem cells from a person called a "donor." The stem cells can be obtained from the hollow part of the hip bone or from blood.

A serious problem with this treatment is graft-versus-host disease (GVHD). This happens when stem cells from the donor attack normal cells of the recipient. Currently, there is no universal standard of care in the United States to prevent GVHD.

This study is being done to see if a medicine that is used to lower cholesterol can also help in reducing GVHD.

Patients will receive atorvastatin daily by mouth starting 14 days before stem cell transplant. They will continue to take atorvastatin until 180 days after transplant. This medicine may be stopped earlier if there is a bad side effect or a severe GVHD. Patients will also receive standard treatment to prevent GVHD. Patients will undergo many tests that are standard for their treatment at West Virginia University (WVU), including blood tests to check blood counts, kidney function and HIV status; blood test to check for pregnancy; Multi Gated Acquisition Scan (MUGA scan)or echocardiogram to test heart function; lung function testing; and bone marrow aspirate or biopsy. Patients will also have the option to provide blood samples for optional research related to the study.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (GVHD) is one of the most frequent complications after allogeneic hematopoietic stem cell transplantation (HSCT).(1) It develops in 30-75% of recipients of allogeneic HSCT depending on the degree of histocompatibility between the donor and the recipient, number of T-cells in the graft, recipient's age and GVHD prophylactic regimen used. (2-4) Novel strategies designed to effectively prevent the development of this life threatening complication of allogeneic transplantation are urgently needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of a hematological malignancy or bone marrow failure syndrome suitable for allogeneic stem cell transplantation in the opinion of treating transplant physician.
* Patients aged 18-75 years of age are eligible. Patients with age > 18 and ≤ 50 years will be eligible for myeloablative conditioning (MAC), while patients > 50 years of age, or those with previous history of autologous transplantation, high hematopoietic cell transplant comorbidity index (HCT-CI) score (>2), and baseline diagnosis of hodgkin's lymphoma, chronic lymphocytic leukemia and follicular lymphoma will be suitable for reduced intensity conditioning (RIC) transplantation (however intensity of conditioning regimen will remain at the discretion of treating physician).
* All patients must have at least one suitable human leukocyte antigen (HLA)-matched sibling or unrelated donor according to transplant center's guidelines (for selection of appropriate sibling donor).
* Patient must provide informed consent.
* Left ventricular ejection fraction ≥ 40%.
* Bilirubin ≤ 2 x the upper limit of normal (ULN) and aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 3 x ULN; and absence of hepatic cirrhosis. For patients with Gilbert's syndrome, bilirubin ≤ 3 x ULN is permitted.
* Adequate renal function as defined by a serum creatinine clearance of ≥ 40% of normal calculated by Cockcroft-Gault equation.
* Carbon monoxide diffusing capacity (DLCOcor) corrected for hemoglobin or forced expiratory volume at one second (FEV1) or DL/VA ≥ 40% of predicted (a pulmonary function test).
* Karnofsky performance status > 70.
* A negative pregnancy test will be required for all women of child bearing potential. Breast feeding is not permitted.
* Patients with positive HIV serology are eligible.
* Patients who have previously been taking atorvastatin or any other statin drug will be eligible as long as there is no contraindication to switch to atorvastatin (40mg/day) in the opinion of the treating physician.
* Method of stem-cell collection from the sibling donor will be at the discretion of the treating physician. Although it is anticipated that majority of sibling donors will undergo Granulocyte colony-stimulating factor(G-CSF) induced stem cell mobilization; however donors undergoing bone marrow harvest or stem cell mobilization with experimental agents (e.g. plerixafor) will remain eligible for the study.

Exclusion Criteria:

* Uncontrolled arrhythmias or uncontrolled New York Heart Association class III-IV heart failure.
* Evidence of active bacterial, viral or fungal infection at the time of transplant conditioning.
* History of intolerance or allergic reactions with atorvastatin will not be eligible.
* Undergoing a T-cell depleted allogeneic transplantation
* Receiving conditioning regimens containing anti-thymocyte globulin, and/or campath

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Craig, MD, Principal Investigator — West Virginia University; Mehdi Hamadani, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deeg HJ. How I treat refractory acute GVHD. Blood. 2007 May 15;109(10):4119-26. doi: 10.1182/blood-2006-12-041889. Epub 2007 Jan 18. PMID 17234737
- [Background] Ratanatharathorn V, Nash RA, Przepiorka D, Devine SM, Klein JL, Weisdorf D, Fay JW, Nademanee A, Antin JH, Christiansen NP, van der Jagt R, Herzig RH, Litzow MR, Wolff SN, Longo WL, Petersen FB, Karanes C, Avalos B, Storb R, Buell DN, Maher RM, Fitzsimmons WE, Wingard JR. Phase III study comparing methotrexate and tacrolimus (prograf, FK506) with methotrexate and cyclosporine for graft-versus-host disease prophylaxis after HLA-identical sibling bone marrow transplantation. Blood. 1998 Oct 1;92(7):2303-14. PMID 9746768
- [Background] Nash RA, Antin JH, Karanes C, Fay JW, Avalos BR, Yeager AM, Przepiorka D, Davies S, Petersen FB, Bartels P, Buell D, Fitzsimmons W, Anasetti C, Storb R, Ratanatharathorn V. Phase 3 study comparing methotrexate and tacrolimus with methotrexate and cyclosporine for prophylaxis of acute graft-versus-host disease after marrow transplantation from unrelated donors. Blood. 2000 Sep 15;96(6):2062-8. PMID 10979948
- [Background] Antin JH, Kim HT, Cutler C, Ho VT, Lee SJ, Miklos DB, Hochberg EP, Wu CJ, Alyea EP, Soiffer RJ. Sirolimus, tacrolimus, and low-dose methotrexate for graft-versus-host disease prophylaxis in mismatched related donor or unrelated donor transplantation. Blood. 2003 Sep 1;102(5):1601-5. doi: 10.1182/blood-2003-02-0489. Epub 2003 May 1. PMID 12730113
- [Background] Liao JK, Laufs U. Pleiotropic effects of statins. Annu Rev Pharmacol Toxicol. 2005;45:89-118. doi: 10.1146/annurev.pharmtox.45.120403.095748. PMID 15822172
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Result] Kanate AS, Hari PN, Pasquini MC, Visotcky A, Ahn KW, Boyd J, Guru Murthy GS, Rizzo JD, Saber W, Drobyski W, Michaelis L, Atallah E, Carlson KS, D'Souza A, Fenske TS, Cumpston A, Bunner P, Craig M, Horowitz MM, Hamadani M. Recipient Immune Modulation with Atorvastatin for Acute Graft-versus-Host Disease Prophylaxis after Allogeneic Transplantation. Biol Blood Marrow Transplant. 2017 Aug;23(8):1295-1302. doi: 10.1016/j.bbmt.2017.04.009. Epub 2017 Apr 12. PMID 28412518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 subjects signed consent. Six did not meet eligibility criteria and were not treated.
Groups:
- Matched Related Donor; Matched Unrelated Donor: Atorvastatin will be administered at a dose of 40 mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning.
  Patients will receive atorvastatin until +180 days or until the patient develops grade II-IV acute GVHD, extensive chronic GVHD, or any grade 3-4 toxicity related to atorvastatin.
  Atorvastatin calcium: 40 mg PO daily
Period: Overall Study
Arm/Group | Matched Related Donor | Matched Unrelated Donor
Started | 30 | 39
Completed | 30 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin Calcium (Lipitor); Unrelated Donor: Atorvastatin will be administered at a dose of 40 mg orally daily starting on day -14, to permit an approximately 1-week observation period to rule out any acute atorvastatin-induced side effects before the initiation of transplant conditioning.
  Patients will receive atorvastatin until +180 days or until the patient develops grade II-IV acute GVHD, extensive chronic GVHD, or any grade 3-4 toxicity related to atorvastatin.
  Atorvastatin calcium: 40 mg PO daily
- Total: Total of all reporting groups
Arm/Group | Atorvastatin Calcium (Lipitor) | Unrelated Donor | Total
Number analyzed (Participants) | 30 | 39 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 29 | 50
  >=65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 17 | 27 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 39 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 28 | 38 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 39 | 69

OUTCOME MEASURES:

1. Primary Outcome: Matched Related Transplants Who Develop Grade II-IV Acute Graft Versus Host Disease (GVHD).
Description: The number of subjects in the matched sibling cohort who develop grades II-IV acute GVHD will be assessed by consensus criteria and graded on Bone Marrow Transplant Clinical Trials Network Manual of Procedures suggested grading sheets. Grade I is mild GVHD involving up to 25% of the subject's skin; Grade II is moderate GVHD. involving 25 to 50% of the subject's skin and can include mild changes in liver and/or mild diarrhea; Grade III is severe GVHD involving over 50% of the subject's skin. Liver involvement is likely as are stomach cramps and diarrhea; and Grade 4 is very severe GvHD. Skin may be blistered and may have broken down in places. Skin may be yellow due to liver injury. Severe diarrhea is common. Subjects in the matched unrelated donors are not included in this analysis.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Related Donor
Number analyzed (Participants) | 30
Participants | 3

2. Primary Outcome: Matched Unrelated Donors Transplants Who Develop Grade II-IV Acute GVHD.
Description: The number of subjects in the matched unrelated donor cohort who develop grade II-IV acute GVHD. Acute GVHD will be assessed by consensus criteria and graded on Bone Marrow Transplant Clinical Trials Network Manual of Procedures suggested grading sheets. Grade I is mild GVHD involving up to 25% of the subject's skin; Grade II is moderate GVHD. involving 25 to 50% of the subject's skin and can include mild changes in liver and/or mild diarrhea; Grade III is severe GVHD involving over 50% of the subject's skin. Liver involvement is likely as are stomach cramps and diarrhea; and Grade 4 is very severe GvHD. Skin may be blistered and may have broken down in places. Skin may be yellow due to liver injury. Severe diarrhea is common. Subjects in the matched related donors are not included in this analysis.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Unrelated Donor
Number analyzed (Participants) | 39
Participants | 12

3. Secondary Outcome: Matched Related Transplants Who Develop Grade II-IV Chronic GVHD.
Description: The number of subjects who develop grade II-IV chronic GVHD. Chronic GVHD diagnosis and grading I to IV will be according to National Institutes of Health (NIH) Criteria rating progressively intense symptoms involving: skin (asymptomatic to deep sclerosis, impaired mobility, ulceration, or pruritus), oral cavity (asymptomatic to symptoms limiting oral intake), eyes (asymptomatic to severe dry eye, inability to work, or loss of vision due to keratoconjunctivitis), gastrointestinal tract (asymptomatic to significant weight loss [>15%] or esophageal dilation), liver (normal function to bilirubin or enzymes >5 times ULN), lungs (asymptomatic to severe shortness of breath requiring supplemental oxygen), joints and fascia (asymptomatic to contractures with reduced range of motion and limited ability to perform daily care), and genital tract (asymptomatic to strictures and severe pain). Subjects in the matched unrelated donors are not included in this analysis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Related Donor
Number analyzed (Participants) | 30
Participants | 9

4. Secondary Outcome: Matched Unrelated Donors Transplants Who Develop Grade II-IV Chronic GVHD.
Description: The number of subjects who develop grade II-IV chronic GVHD. Chronic GVHD diagnosis and grading I to IV will be according to National Institutes of Health (NIH) Criteria rating progressively intense symptoms involving: skin (asymptomatic to deep sclerosis, impaired mobility, ulceration, or pruritus), oral cavity (asymptomatic to symptoms limiting oral intake), eyes (asymptomatic to severe dry eye, inability to work, or loss of vision due to keratoconjunctivitis), gastrointestinal tract (asymptomatic to significant weight loss [>15%] or esophageal dilation), liver (normal function to bilirubin or enzymes >5 times ULN), lungs (asymptomatic to severe shortness of breath requiring supplemental oxygen), joints and fascia (asymptomatic to contractures with reduced range of motion and limited ability to perform daily care), and genital tract (asymptomatic to strictures and severe pain). Subjects in the matched related donors are not included.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Unrelated Donor
Number analyzed (Participants) | 39
Participants | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Atorvastatin Calcium (Lipitor) | Unrelated Donor
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/39
Serious Adverse Events (participants affected / at risk) | 10/30 | 12/39
Other Adverse Events (participants affected / at risk) | 30/30 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin Calcium (Lipitor) (N=30) | Unrelated Donor (N=39)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Bilirubin increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin Calcium (Lipitor) (N=30) | Unrelated Donor (N=39)
Anemia (Blood and lymphatic system disorders) | 13 (18) | 23 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 9 (9)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (2) — Carotid artery disease
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Neck lesion biopsy
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Pollen allergy (Immune system disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Scabies (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 4 (4)
Multiple drug resistant infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 5 (5) | 7 (7)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 8 (8)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Transfusion reaction
Alanine aminotransferase increased (Investigations) | 5 (7) | 4 (7)
Alkaline phosphatase increased (Investigations) | 3 (3) | 5 (6)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Cholesterol high (Investigations) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Dyslipidemia (Investigations) | 1 (1) | 0 (0)
Ferritin increased (Investigations) | 1 (3) | 4 (4)
Lactate dehydrogenase increased (Investigations) | 4 (4) | 7 (7)
Red blood cell count decreased (Investigations) | 11 (11) | 11 (11)
Chloride increased (Investigations) | 5 (5) | 4 (4)
Blood urea nitrogen increased (Investigations) | 1 (1) | 1 (1)
Total protein decreased (Investigations) | 1 (1) | 6 (6)
Lactate dehydrogenase decreased (Investigations) | 0 (0) | 3 (3)
Hematocrit decreased (Investigations) | 0 (0) | 1 (1)
Hypercholesterolemia (Investigations) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 2 (2)
Monocyte count increased (Investigations) | 1 (1) | 2 (2)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0)
Chloride decreased (Investigations) | 1 (1) | 0 (0)
Bicarbonate decreased (Investigations) | 1 (1) | 1 (1)
Blood Urea Nitrogen decreased (Investigations) | 1 (1) | 0 (0)
Eosinophils decreased (Investigations) | 0 (0) | 1 (1)
Anion gap high (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase decreased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 15 (15) | 14 (14)
Neutrophil count decreased (Investigations) | 17 (17) | 17 (17)
Platelet count decreased (Investigations) | 14 (14) | 15 (15)
Anorexia (Metabolism and nutrition disorders) | 15 (15) | 17 (17)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10) | 12 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Drug-induced myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Uterine polyps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 3 (3)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Breast infection (Infections and infestations) | 1 (1) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic occlusive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Appendectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Cholesystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac stent placed (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Nissen fundoplication (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin grafts trunk arm leg 100 cm^2 or less (Surgical and medical procedures) | 0 (0) | 1 (1)
Inferior vena cava filter placed (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 10 (11)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 5 (5)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT01665677/Prot_SAP_000.pdf
  • Informed Consent Form (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT01665677/ICF_001.pdf